CLINICAL TRIAL: NCT04813172
Title: The Implementation of Enhanced Care Coordination in Order to Decrease Hospital Utilization for Head & Neck Survivors Undergoing Radiation
Brief Title: Enhanced Care Coordination for Head and Neck Cancer Survivors
Acronym: ECC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Marci Nilsen, Assistant Professor Acute & Tertiary Care, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY19120089
Record Dates: First submitted 2021-03-01; First posted 2021-03-24 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Head and neck cancer patients (Experimental): Patients from the Eye and Ear Institute Survivorship Clinic who are diagnosed with head and neck cancer.
  Interventions: Behavioral: Symptom Assessment

INTERVENTIONS:
Behavioral: Symptom Assessment — Examine the symptomatology of head and neck cancer patients undergoing treatment that includes radiation by completing the M.D. Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN), the Brief Pain Index (BPI)and the Functional Assessment of Cancer Therapy for Head and Neck Cancer (FACT-H&N). They will also be asked to complete the Hearing Handicap Inventory for Adults - Screening (HHIA-S) and the Tinnitus Handicap Inventory - Screening (THI-S) as well as the Flourishing Measure.
  Each patient enrolled will be followed by a nurse and speech-language pathologist, twice a week, throughout their treatment (from start until 3-month post completion) All assessments are collected on a secure Ipad through REDcap database. If any significant changes occur, within 2 points from their last assessment, the nurse will notify the oncology physician and provide plan of care to avoid emergency room or hospital visit.

SUMMARY:
The purpose of this study is to evaluate the effect of a multidimensional symptom management intervention on decreasing symptom burden and thus reducing hospital utilization in patients undergoing radiation with or without chemotherapy for head and neck cancer.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of a multidimensional symptom assessment intervention on identifying symptoms and alerting care team of changes, and thus reducing hospital utilization, in patients undergoing radiation with or without chemotherapy for head and neck cancer. This is a pilot study.

This project is being conducted to 1) examine the symptomatology of head and neck cancer patients undergoing treatment that includes radiation, 2) determine the hospital admission rates of this patient population before, during and post treatment, 3) compare the admission rates of this patient population to historical controls and 4) to examine overall patient compliance.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Diagnosed with primary, head and neck cancer of the paranasal sinuses, nasal cavity, oral cavity, tongue, salivary glands, larynx, and pharynx (including the nasopharynx, oropharynx, and hypopharynx)
* Will include squamous cell carcinoma found in lymph nodes as a result of unknown primary location.
* Prior to the initiation of radiation treatment for qualifying diagnosis
* Treatment occurring at Hillman Cancer Center

Exclusion Criteria:

* Prior radiation treatment of squamous cell carcinoma of the locations listed in inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Emergency Room Visits | Start of treatment to 3 month post treatment completion
  The total number number of emergency room visits from start of radiation therapy until 90 days after treatment completion.
Inpatient Hospitalizations | Start of treatment to 3 month post treatment completion
  The total number number of inpatient hospital from start of radiation therapy until 90 days after treatment completion.. The length of each stay will also be counted by the number of days.

SECONDARY OUTCOMES:
M.D. Anderson Symptom Inventory for Head and Neck Cancer | Start of treatment to 3 month post treatment completion
  The M.D. Anderson Symptom Inventory for Head and neck Cancer is to assess the severity of symptoms experienced by patients with cancer and the interference with daily living caused by these symptoms.
  It uses a 0-10 scale "0" (the symptom was "NOT present") to "10" (the symptom was "As bad as you can imagine"). Higher score is worse outcome.
Brief Pain Index (BPI) | Start of treatment to 3 month post treatment completion
  The Brief Pain Inventory (BPI) rapidly assesses the severity of pain and its impact on functioning in the past 24 hours.
  It uses a 0-10 scale "0" (the symptom was "NOT present") to "10" (the symptom was "As bad as you can imagine").
  The higher the score is worse outcome.
Functional Assessment of Cancer Therapy for Head and Neck Cancer | Start of treatment to 3 month post treatment completion
  The Functional Assessment of Cancer Therapy for Head and neck Cancer assesses 5 domains Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being over the past 7 days.
  It uses a 5 point Likert Scale: Not at all, A little bit, Somewhat, Quite a bit, Very much to rate functioning in the 5 domains.
  The higher the score, the better the outcome/quality of life.
Hearing Handicap Inventory for Adults | Start of treatment to 3 month post treatment completion
  This self-assessment tool is designed to assess the effects of hearing loss and impairment while going through radiation treatment.
  It is a 10 item instrument that patients select YES, SOMETIMES or NO for each question.
  A total possible score ranges from minimum score of 0 to maximum score of 40.
  The higher the score, the more handicap they have due to hearing loss and impairment.
Tinnitus Handicap Inventory | Start of treatment to 3 month post treatment completion
  This self assessment tool is designed to assess the severity of tinnitus handicap as well as predicting the psychological distress associated with tinnitus. The instrument consist of three subscales comprising 4 emotional items ,4 functional items and 2 catastrophic items.
  It is a 10 item instrument that patients select YES, SOMETIMES or NO for each question. A total possible score ranges from minimum score of 0 to maximum score of 40.
  The higher the score, the more handicap they have due to tinnitus.
Flourishing Measure | Start of treatment to 3 month post treatment completion
  The Flourishing Scale is a brief 10-item summary measure of the respondent's self-perceived success in important areas such as relationships, self-esteem, purpose, and optimism. The scale provides a single psychological well-being score.
  Minimum score is 0 (not satisfied) and maximum score is 10 (extremely satisfied)
  A high score represents a person with many psychological resources and strengths. A low score represents a person with limited psychological resources and limitations.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye and Ear Institute, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No